CLINICAL TRIAL: NCT02470065
Title: Resectable EGFR Mutant NSCLC With (or Without) Afatinib as Neoadjuvant Treatment; REMNANT an Exploratory Study of the EORTC Lung Cancer Group
Brief Title: Neoadjuvant Afatinib in Early Stage Non Small Cell Lung Cancer.
Acronym: REMNANT
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-08115
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Early stage; Phase II; Randomized; EGFR mutated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neo adjuvant afatinib (Experimental): once daily afatinib at a dose of 40 mg for 8 weeks followed by surgery with curative intent (anatomical resection and systematic lymph node dissection).
  Interventions: Drug: Afatinib; Procedure: Immediate surgery
- Immediate surgery (Active Comparator): immediate surgery with curative intent (anatomical resection and systematic lymph node dissection).
  Interventions: Procedure: Immediate surgery

INTERVENTIONS:
Drug: Afatinib — once daily afatinib at a dose of 40 mg for 8 weeks
  Arms: Neo adjuvant afatinib
Procedure: Immediate surgery — anatomical resection and systematic lymph node dissection

SUMMARY:
This is a multicenter, randomized, 1:1, non-comparative phase II trial. Patients with early stage NSCLC will be randomized between ARM A: neoadjuvant afatinib followed by surgery and ARM B: immediate surgery with curative intent.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, randomized, non-comparative, two-arm phase II trial aiming to evaluate afatinib treatment in pre-operative setting in patients with EGFR mutated NSCLC.

After signing of the informed consent, patients will be registered and screened for eligibility and upon confirmation of all eligibility criteria, patients will be randomized 1:1 to:

* Arm A: once daily afatinib at a dose of 40 mg for 8 weeks followed by surgery with curative intent (anatomical resection and systematic lymph node dissection).
* Arm B: immediate surgery with curative intent (anatomical resection and systematic lymph node dissection).

Response evaluation in the pre-operative arm will be performed through CT scans at baseline, 4 and 8 weeks.

The first 5 patients enrolled in arm A will be part of a safety run-in to check that afatinib treatment doesn't delay surgery.

ELIGIBILITY:
Inclusion Criteria:

Histological or cytological diagnosis of NSCLC;

* Patients considered operable and with resectable tumor with curative intent (anatomical resection and systematic lymph node dissection) based on evaluation by a thoracic multi-disciplinary team composed of at least a thoracic surgeon, oncologist and radiologist;
* Stage I-III (T1a-3, N0-1, M0 according to UICC version 7) NSCLC by local staging criteria potentially treatable by radical (curative) surgery. Patients with T1 tumor at baseline will be limited to 20%;
* Radiologically measurable disease according to RECIST criteria 1.1; assessed by chest and upper abdomen CT scan within 2 weeks (+1 week) prior to registration); brain CT scan or MRI according to local practice;
* No prior treatment for NSCLC is allowed;
* Adequate tissue in terms of quality and quantity for EGFR local testing.

Exclusion Criteria:

* no adequate bone marrow function within 2 weeks prior to randomization
* no adequate liver function. Patients with Gilbert's syndrome total bilirubin must be below 4 times institutional upper limit of normal; within 2 weeks prior to randomization
* no adequate renal function within 2 weeks prior to randomization
* known positivity to human immunodeficiency virus (HIV), hepatitis B or hepatitis C;
* known history of allergic reactions attributed to compounds of similar chemical or biological composition;
* history of a hematologic or primary solid tumor malignancy, unless no evidence of that disease for 5 years, except pT1-2 prostatic cancer Gleason score < 6, superficial bladder cancer, non melanoma skin cancer or carcinoma in situ of the cervix;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-09 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in cT-stage | 8 weeks
  decrease in cT-stage descriptor measured according to RECIST 1.1

SECONDARY OUTCOMES:
Response Rate | 8 weeks
  proportion of patients whose response is either complete response (CR) or partial response (PR) using RECIST 1.1;
Change in surgical treatment intent and technique | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Popat, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust